CLINICAL TRIAL: NCT06104618
Title: Phase II Study of Enfortumab Vedotin Treatment for Metastatic Squamous Cell Carcinoma of the Penis
Brief Title: Enfortumab Vedotin for the Treatment of Patients With Metastatic or Unresectable Squamous Cell Carcinoma of the Penis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC200505; NCI-2023-08624 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 20-011329 (Other: Mayo Clinic Institutional Review Board); MC200505 (Other: Mayo Clinic in Rochester)
Record Dates: First submitted 2023-10-23; First posted 2023-10-27 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Metastatic Penile Squamous Cell Carcinoma; Stage III Penile Cancer AJCC v8; Stage IV Penile Cancer AJCC v8; Unresectable Penile Squamous Cell Carcinoma
MeSH Terms: conditions — Penile Neoplasms | interventions — enfortumab vedotin; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (Enfortumab vedotin) (Experimental): Patients receive enfortumab vedotin IV over 30 minutes on days 1,8 and 15 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo CT or MRI throughout the study.
  Interventions: Drug: Enfortumab Vedotin; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging

INTERVENTIONS:
Drug: Enfortumab Vedotin — Given IV
  Other Names: AGS 22ME; AGS-22M6E; Anti-Nectin 4 ADC ASG-22CE; Anti-nectin-4 Monoclonal Antibody-Drug Conjugate AGS-22M6E; ASG-22CE; Enfortumab Vedotin-ejfv; Padcev
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; computerized axial tomography; Computerized Axial Tomorgraphy; computed axial tomogrpahy; Computerized Tomography; computerized tmography; Computerized Tomography (CT) scan; CT; CT Scan
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: MRI; Magnetic Resonance Imaging (MRI); Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MRI Scan; NMR Imaging; NMRI; nuclear magnetic resonance imaging; Nuclear Resonance Magnetic Imaging; structural MRI; sMRI

SUMMARY:
This phase II trial tests how well enfortumab vedotin works for treating patients with squamous cell carcinoma of the penis that has spread to other places in the body (metastatic) or cannot be removed by surgery (unresectable). Enfortumab vedotin is a monoclonal antibody, enfortumab, linked to an anticancer drug called vedotin. It works by helping the immune system to slow or stop the growth of tumor cells. Enfortumab attaches to a protein called nectin-4 on tumor cells in a targeted way and delivers vedotin to kill them.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To estimate the best response rate of enfortumab vedotin treatment for patients with metastatic penile squamous cell carcinoma (mPSCC).

SECONDARY OBJECTIVES:

I. To determine overall response rate (ORR). II. To determine safety and tolerance of enfortumab vedotin in men with mPSCC. III. To characterize duration of response to enfortumab vedotin in mPSCC. IV. To estimate median overall survival and progression-free survival in men with mPSCC treated with enfortumab vedotin.

V. To analyze response in subgroups by human papillomavirus (HPV) status (related/unrelated as assessed by p16 biomarker).

OUTLINE:

Patients receive enfortumab vedotin intravenously (IV) over 30 minutes on days 1,8 and 15 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo computed tomography (CT) or magnetic resonance imaging (MRI) throughout the study.

After completion of study treatment, patients are followed up at 30 days and then every 3 months until progressive disease, followed by every 6 months for up to 5 years from registration.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Histological confirmation of squamous cell carcinoma of the penis (PSCC): NOTE: Biopsy confirmation of at least one site of metastasis is encouraged but not required.
* At least one site of metastatic or unresectable PSCC. NOTE: Prior therapy is not required for patients whose treatment is considered palliative (for example, presence of distant metastasis). NOTE: Patients who are potentially curable (any T, N1 - N3, M0) must have had tumor progression after standard chemotherapy, radiotherapy, or surgery, or be unable to receive such treatment. Eligible stages include:

  * Any T, N1 (i.e., a palpable mobile unilateral inguinal lymph node), M0 OR
  * Any T, N2 (i.e., palpable mobile multiple or bilateral inguinal lymph nodes), M0 OR
  * Any T, N3 (i.e., fixed inguinal nodal mass or any pelvic lymphadenopathy), M0 OR
  * Any T, any N, M1
* Patients with clinical N1, M0 mPSCC at protocol entry must be ineligible for surgery because of comorbidities or clinical T4 disease, or have refused surgery
* Patients with clinical N1 - N3, M0, and no prior systemic therapy must be:

  * Unable to receive neoadjuvant (paclitaxel + ifosfamide + cisplatin) TIP because of comorbidities or refused TIP; AND
  * Unable to receive radiotherapy with curative intent, or refused radiotherapy
* Measurable disease by Response Evaluation Criteria in Solid Tumors (RECIST 1.1)
* Prior therapy is allowed. Patients may be treatment-naïve or have had any number of prior anti-cancer treatments
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0 or 1
* Hemoglobin ≥ 9.0 g/dL obtained ≤15 days prior to registration
* Absolute neutrophil count (ANC) ≥ 1000/mm^3 obtained ≤ 15 days prior to registration
* Platelet count ≥ 100,000/mm^3 obtained ≤ 15 days prior to registration
* Total bilirubin ≤ 1.5 x upper limit of normal (ULN) or ≤ 3 x ULN for patients with Gilbert's disease obtained ≤ 15 days prior to registration
* Alanine aminotransferase (ALT) and aspartate transaminase (AST) ≤ 2.5 x ULN obtained ≤ 15 days prior to registration
* Glomerular filtration rate (GFR) or calculated creatinine clearance ≥ 30 ml/min as estimated using the Cockcroft-Gault formula or as measured by 24-hour urine collection obtained ≤ 15 days prior to registration
* Provide written informed consent
* Willing to return to enrolling institution for follow-up (during the active monitoring phase of the study)

Exclusion Criteria:

* Pure verrucous carcinoma of the penis
* Non-squamous malignancy of the penis
* Squamous carcinoma of the urethra
* Preexisting sensory or motor neuropathy ≥ grade 2
* Active central nervous system (CNS) metastases. Exception: Treated CNS metastases are allowed if all of the following are true:

  * CNS metastases are clinically stable for ≥ 6 weeks prior to registration
  * If needed, steroid dose is stable and ≤ 20 mg/day of prednisone or equivalent for ≥ 2 weeks prior to registration
  * Baseline imaging shows no evidence of new or enlarged brain metastasis
  * No leptomeningeal disease
* History of uncontrolled diabetes mellitus ≤ 3 months prior to registration NOTE: Uncontrolled diabetes is defined as hemoglobin A1c (HbA1c) ≥ 8.0% or HbA1c 7.0-7.9% with associated diabetes symptoms (polyuria or polydipsia) that are not otherwise explained
* Failure to recover from any of the following therapies prior to registration:

  * Major surgery
  * Radiotherapy, chemotherapy, biologics, investigational agents, and/or antitumor treatment with immunotherapy
* Immunocompromised patients and patients known to be human immunodeficiency virus (HIV) positive
* Uncontrolled intercurrent illness including, but not limited to:

  * Ongoing or active infection requiring systemic treatment
  * History of cerebral vascular event (stroke or transient ischemic attack)
  * Myocardial infarction or symptomatic congestive heart failure (New York Heart Association [NYHA] Class III-IV) ≤ 6 months prior to registration
  * Unstable angina pectoris
  * Cardiac arrhythmia
  * Or psychiatric illness/social situations that would limit compliance with study requirements (e.g., history of substance abuse)
* Receiving any other investigational agent which would be considered as a treatment for the primary neoplasm
* Currently receiving systemic antimicrobial treatment for viral, bacterial or fungal infection. NOTE: Routine antimicrobial prophylaxis is allowed
* Known active hepatitis B (e.g., hepatitis B surface antigen [HBsAg] reactive) or active hepatitis C (e.g., hepatitis C virus [HCV] ribonucleic acid (RNA) [qualitative] is detected)
* Known active keratitis or corneal ulcerations. NOTE: Superficial punctate keratitis is allowed if the disorder is being adequately treated
* Known hypersensitivity to enfortumab vedotin or to any excipient contained in the drug formulation of enfortumab vedotin (including histidine, trehalose dihydrate and polysorbate 20) OR subject has known hypersensitivity to biopharmaceutical produced in Chinese hamster ovary cells
* Other active malignancy ≤ 2 years prior to registration. EXCEPTIONS: Locally curable cancers that have been apparently cured such as basal or squamous cell skin cancer, non-muscle-invasive bladder cancer, or carcinoma in situ of the breast or low risk Gleason 6 prostate cancer.
* History of myocardial infarction ≤ 6 months, or congestive heart failure requiring use of ongoing maintenance therapy for life-threatening ventricular arrhythmias
* Patients who are sexually active and unwilling to use effective contraception (if they are not already surgically sterile)
* Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens
* Chemotherapy-naïve patients who are potentially curable (any T, N1 - N3, M0) in the absence of any condition that precludes cisplatin-based chemotherapy, such as low GFR, peripheral neuropathy, hearing impairment, or psychosocial considerations

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2023-12-21 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Best response rate | Up to 5 years
  Defined as the proportion of patients who experience either a partial response (PR) or complete response (CR) as defined by Response Evaluation Criteria in Solid Tumors (RECIST) version (v) 1.1. The best response rate of CR/PR will be reported descriptively and a 95% confidence interval will be reported.

SECONDARY OUTCOMES:
Objective response rate (ORR) | Up to 5 years
  Defined as the proportion of patients who experience either a confirmed partial response or confirmed complete response as defined by RECIST v1.1. ORR will be reported descriptively and a 95% confidence interval will be reported.
Progression free survival (PFS) | From study entry to the first of either disease progression or death from any cause, up to 5 years
  Will be estimated using the Kaplan-Meier method. The median PFS and 95% confidence interval will be reported.
Overall survival (OS) | From study entry to death from any cause, up to 5 years
  Will be estimated using the Kaplan-Meier method. The median OS and 95% confidence interval will be reported.
Incidence of adverse events | Up to 30 days after last dose of study medication
  The maximum grade for each type of adverse event by patient will be summarized by frequencies and percentages using Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
Duration of Response | Up to 5 years
  Defined for all evaluable patients who have achieved an objective response as the date at which the patient's earliest best objective status is first noted to be either a CR or PR to the earliest date progression is documented.
Best response by human papillomavirus (HPV) status | Up to 5 years
  The p16 biomarker will be used to assess HPV status. The p16 immunohistochemistry (IHC) outcome will be classified as positive, negative, or not available. Best response rates of either a CR or PR will be determined for each subgroup and 95% confidence intervals will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Lance C. Pagliaro, M.D., Principal Investigator — Mayo Clinic in Rochester
Locations (3):
- United States (3):
  - Mayo Clinic Hospital in Arizona, Phoenix, Arizona
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Mayo Clinic in Rochester, Rochester, Minnesota

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials